CLINICAL TRIAL: NCT04657263
Title: Impact of the COVID-19 Pandemic on Vaccination in Patients at Risk of Infection
Brief Title: Impact of the COVID-19 Pandemic on Vaccination
Acronym: COVIDVacImpac
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0655
Record Dates: First submitted 2020-12-07; First posted 2020-12-08 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Covid19
Keywords: People over 18 years old; vaccines; immunization schedule; Infection
MeSH Terms: conditions — COVID-19; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Person at risk of infection according to French 2019 immunization: Person at risk of infection according to French 2019 immunization
  Interventions: Other: Vaccine coverage assessment

INTERVENTIONS:
Other: Vaccine coverage assessment — Vaccine coverage assessment

SUMMARY:
The vaccination policy is drawn up in France by the French Minister of Health, who makes public the vaccination schedule after the opinion of the High Authority of Health.

Currently according to the 2019 immunization schedule, the dTP vaccine is the only mandatory in the general population with recalls in adults aged 25, 45, 65 and every 10 years. In 2011, the Ministry of Health estimated that only 50.5% of the general population was up to date against dTP.

Two vaccines are recommended for person at risk of infection according to the current vaccine schedule: the flu vaccine and the pneumococcal vaccine. In fact, influenza and pneumococcal disease are more frequent and more serious in patients with chronic diseases (diabetes, cardiac insufficiency..) compared to the general population.

The vaccination coverage rate of at-risk populations is dramatically below the vaccination coverage targets set by the Ministry of Health. Indeed, there are many barriers to vaccination, medical and para-medical barriers, but also individual barriers.

The current COVID-19 pandemic has identified people at risk of severe infection and death risk, particularly those with co-morbidities (diabetes, cardiovascular disease, etc.). Thus, this pandemic may have contributed to change in patients' perceptions regarding both the risk of infection and the potential interest and benefit of vaccination.

ELIGIBILITY:
Inclusion criteria:

* Person at risk of infection according to french 2019 immunization schedule
* Patients aged above 18 years old

Exclusion criteria:

- Patient < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was composed of person at risk of infection cared for in participating centers
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
number of persons at risk of infection up to date with their mandatory and recommended vaccinations during COVID19 pandemic | 1 day
  number of persons at risk of infection up to date with their mandatory and recommended vaccinations during COVID19 pandemic

SECONDARY OUTCOMES:
Number of persons at risk of infection accepting COVID19 vaccination | 1 day
  Number of persons at risk of infection accepting COVID19 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Cyril BREUKER, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC